CLINICAL TRIAL: NCT02881320
Title: A Phase 2/3, Open-Label Study of the Pharmacokinetics, Safety, and Antiviral Activity of the GS-9883/Emtricitabine/Tenofovir Alafenamide (GS-9883/F/TAF) Fixed Dose Combination (FDC) in HIV-1 Infected Adolescents and Children
Brief Title: Study of Bictegravir/Emtricitabine/Tenofovir Alafenamide Fixed Dose Combination in Adolescents and Children With Human Immunodeficiency Virus-1
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-380-1474; 2016-002345-39 (EudraCT Number)
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 (12 to < 18 years of age and weight ≥ 35 kg) (Experimental): * Part A: Participants will participate in an Intensive PK evaluation at Week 2 or Week 4 and continue to receive the adult strength B/F/TAF FDC through Week 48.
  * Part B: Following confirmation of BIC PK data from Cohort 1 Part A, participants will receive the adult strength B/F/TAF through Week 48.
  Interventions: Drug: B/F/TAF (Adult Strength)
- Cohort 2 (6 to < 12 years of age and weight ≥ 25 kg) (Experimental): * Part A: Participants will participate in an Intensive PK evaluation at Week 2 or Week 4 and continue to receive the adult strength B/F/TAF FDC through Week 48.
  * Part B: Following confirmation of BIC PK data from Cohort 2 Part A, participants will receive the adult strength B/F/TAF FDC through Week 48.
  Interventions: Drug: B/F/TAF (Adult Strength)
- Cohort 3 (≥ 2 years of age and weight ≥ 14 to < 25 kg) (Experimental): * Part A: Participants will participate in an Intensive PK evaluation at Week 2 after which they will continue to receive the low dose B/F/TAF FDC tablet through Week 48.
  * Part B: Following confirmation of BIC PK data from Cohort 3 Part A, participants will receive the low dose B/F/TAF FDC tablet through Week 48.
  Interventions: Drug: B/F/TAF (Low Dose)
- Cohort 4 Group 1 (≥ 2 years of age and weight ≥ 14 to < 25 kg) (Experimental): Due to Cohort 3 Part A Intensive PK evaluation at Week 2 with the low dose B/F/TAF FDC tablet, participants will not participate in an Intensive PK evaluation at Week 2.
  Participants will receive B/F/TAF FDC tablets for oral suspension (TOS) once daily through Week 48.
  Interventions: Drug: B/F/TAF (TOS)
- Cohort 4 Group 2 (≥ 1 month of age and weight ≥ 10 to < 14 kg) (Experimental): Participants will participate in an Intensive PK evaluation at Week 2 after which they will continue to receive B/F/TAF FDC TOS twice daily through Week 48.
  Interventions: Drug: B/F/TAF (TOS)
- Cohort 4 Group 3 (≥ 1 month of age and weight ≥ 6 to < 10 kg) (Experimental): Participants will participate in an Intensive PK evaluation at Week 2 after which they will continue to receive B/F/TAF FDC TOS twice daily through Week 48.
  Interventions: Drug: B/F/TAF (TOS)
- Cohort 4 Group 4 (≥ 1 month of age and weight ≥ 3 to < 6 kg) (Experimental): Participants will participate in an Intensive PK evaluation at Week 2 after which they will continue to receive B/F/TAF FDC TOS twice daily through Week 48.
  Interventions: Drug: B/F/TAF (TOS)
- Open-Label Extension (Experimental): Following Week 48, participants in countries where B/F/TAF is not available may have the option to receive adult strength B/F/TAF FDC, low dose B/F/TAF FDC, or B/F/TAF FDC TOS (based on age and weight) until it becomes available for use according to the participant's age and weight or the product becomes accessible to participants through an access program.
  Interventions: Drug: B/F/TAF (Adult Strength); Drug: B/F/TAF (Low Dose); Drug: B/F/TAF (TOS)

INTERVENTIONS:
Drug: B/F/TAF (Adult Strength) — 50/200/25 mg FDC tablets administered orally once daily without regard to food.
  Other Names: Biktarvy®; GS-9883/F/TAF
  Arms: Cohort 1 (12 to < 18 years of age and weight ≥ 35 kg); Cohort 2 (6 to < 12 years of age and weight ≥ 25 kg); Open-Label Extension
Drug: B/F/TAF (Low Dose) — 30/120/15 mg FDC tablets administered orally once daily without regard to food.
  Other Names: GS-9883/F/TAF
  Arms: Cohort 3 (≥ 2 years of age and weight ≥ 14 to < 25 kg); Open-Label Extension
Drug: B/F/TAF (TOS) — 2 x B/F/TAF 15/60/7.5 mg (total daily dose 30/120/15 mg) FDC tablets administered orally as TOS, once daily.
  Other Names: GS-9883/F/TAF
  Arms: Cohort 4 Group 1 (≥ 2 years of age and weight ≥ 14 to < 25 kg); Open-Label Extension
Drug: B/F/TAF (TOS) — 2 x B/F/TAF 3.75/15/1.88 mg (total daily dose 15/60/7.52 mg) FDC tablets administered orally as TOS, twice daily.
  Other Names: GS-9883/F/TAF
  Arms: Cohort 4 Group 2 (≥ 1 month of age and weight ≥ 10 to < 14 kg); Open-Label Extension
Drug: B/F/TAF (TOS) — 1 x B/F/TAF 3.75/15/1.88 mg (total daily dose 7.5/30/3.76 mg) FDC tablets administered orally as TOS, twice daily.
  Other Names: GS-9883/F/TAF
  Arms: Cohort 4 Group 3 (≥ 1 month of age and weight ≥ 6 to < 10 kg); Open-Label Extension
Drug: B/F/TAF (TOS) — 1 x B/F/TAF 1.88/7.5/0.94 mg (total daily dose 3.76/15/1.88 mg) FDC tablets administered orally as TOS, twice daily
  Other Names: GS-9883/F/TAF
  Arms: Cohort 4 Group 4 (≥ 1 month of age and weight ≥ 3 to < 6 kg); Open-Label Extension

SUMMARY:
The goals of this clinical study are to learn how Bictegravir/Emtricitabine/Tenofovir Alafenamide fixed dose combination (FDC) interacts with the body, confirm the dose, and also to learn more about the safety and tolerability of Bictegravir/Emtricitabine/Tenofovir Alafenamide FDC in adolescents and children with HIV-1.

ELIGIBILITY:
Key Inclusion Criteria:

Cohort 1: HIV-1 infected adolescents (12 to < 18 years of age and screening weight ≥ 35 kg) who are virologically suppressed for ≥ 6 months prior to screening. Cohort 2: HIV-1 infected children (6 to < 12 years of age and screening weight ≥ 25 kg) who are virologically suppressed for ≥ 6 months prior to screening.

Cohort 3: HIV-1 infected children (≥ 2 years of age and screening weight of ≥ 14 to < 25 kg) who are virologically suppressed for ≥ 6 months prior to screening.

Cohort 4 Group 1: HIV-1 infected children (≥ 2 years of age and screening weight of ≥ 14 to < 25 kg) who are virologically suppressed for ≥ 6 months prior to screening and unable to swallow tablets.

* Documented plasma HIV-1 ribonucleic acid (RNA) < 50 copies/mL on a stable regimen (or undetectable HIV-1 RNA level according to the local assay being used if the limit of detection is ≥ 50 copies/mL) for ≥ 6 months preceding the Screening visit. Unconfirmed virologic elevations of ≥ 50 copies/mL (transient detectable viremia, or "blip") prior to screening are acceptable. If the lower limit of detection of the local HIV-1 RNA assay is < 50 copies/mL (eg, < 20 copies/mL), the plasma HIV-1 RNA level cannot exceed 50 copies/mL on two consecutive HIV-1 RNA tests.
* Stable antiretroviral regimen of 2 nucleoside reverse transcriptase inhibitors (NRTIs) in combination with a third agent for a minimum of 6 months prior to the screening visit. Individuals undergoing dose modifications to their antiretroviral regimen for growth or who are switching medication formulation(s) are considered to be on a stable antiretroviral regimen.
* Estimated glomerular filtration rate (eGFR) ≥ 90 mL/min/1.73 m^2 according to the Schwartz Formula.
* No documented or suspected resistance to emtricitabine (FTC), tenofovir (TFV), or integrase strand transfer inhibitors (INSTIs) including, but not limited to, the reverse transcriptase resistance mutations K65R and M184V/I.

Cohort 4 Group 2-4: HIV-1 infected children (≥ 1 month of age and screening weight of ≥ 3 to < 14 kg) who are treatment naive or on antiretroviral (ARV) treatment for ≥ 1 month prior to screening.

* Positive confirmatory HIV test (confirmatory nucleic acid-based testing if < 18 months of age).
* On a stable ARV regimen for ≥ 1 month or treatment naive (Individual is considered treatment naive if ARVs were given for prevention of mother-to-child transmission but not for HIV treatment).
* For < 1 year of age, eGFR ≥ the minimum normal values for age according to the information below using the Schwartz Formula,

  * 30 mL/min/1.73 m^2 for age > 4 weeks to ≤ 95 days.
  * 39 mL/min/1.73 m^2 for age ≥ 96 days to ≤ 6 months.
  * 49 mL/min/1.73 m^2 for age > 6 months to < 12 months.
* For ≥ 1 year of age, eGFR ≥ 90 mL/min/1.73 m^2 using the Schwartz Formula.
* No documented or suspected resistance to FTC, TFV, or INSTIs including, but not limited to, the reverse transcriptase resistance mutation K65R.
* For individuals < 14 kg, M184V/I AND HIV-1 RNA < 50 copies/mL will be allowed. Individuals with HIV-1 RNA > 50 copies/mL should not have FTC, TFV, or INSTI resistance mutations.
* Last dose of nevirapine (NVP) or efavirenz (EFV), if applicable, ≥ 14 days prior to enrollment.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 177 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
PK Parameter: AUCtau of Bictegravir | Week 2 or Week 4 for Cohorts 1 & 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, & 24 hours postdose; Week 2 for Cohort 3: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, & 24 hours post-dose; Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval). Cohorts 1 & 2 Part A will participate in an Intensive PK Evaluation at Week 2 or Week 4. Samples will be collected at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post-dose.
  Cohort 3 Part A will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose.
  Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
PK Parameter: Ctau of Bictegravir | Week 2 or Week 4 for Cohorts 1 & 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, & 24 hours postdose; Week 2 for Cohort 3: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, & 24 hours post-dose; Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  Ctau is defined as the observed drug concentration at the end of the dosing interval. Cohorts 1 & 2 Part A will participate in an Intensive PK Evaluation at Week 2 or Week 4. Samples will be collected at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post-dose.
  Cohort 3 Part A will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose.
  Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
PK Parameter: AUC0-24 of TAF (Cohort 4) | Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  AUClast is defined as area under the concentration versus time curve from time zero to the last quantifiable concentration.
  Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
PK Parameter: AUC0-24 of Bictegravir (Cohort 4) | Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  AUClast is defined as area under the concentration versus time curve from time zero to the last quantifiable concentration.
  Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
PK Parameter: Cmax of TAF (Cohort 4) | Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  Cmax is defined as maximum observed concentration of drug. Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
Percentage of Participants Experiencing Treatment-Emergent Adverse Events (AEs) Through Week 24 | Up to 24 weeks
Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities Through Week 24 | Up to 24 weeks

SECONDARY OUTCOMES:
Proportion of Participants with Plasma HIV-1 RNA < 50 copies/mL at Week 24 as Defined by the US FDA-Defined Snapshot Algorithm | Week 24
Proportion of Participants with Plasma HIV-1 RNA < 50 copies/mL at Week 48 as Defined by the US FDA-Defined Snapshot Algorithm | Week 48
Change from Baseline in CD4+ Cell Counts at Week 24 | Baseline, Week 24
Change from Baseline in CD4+ Cell Counts at Week 48 | Baseline, Week 48
Change from Baseline in CD4+ Cell Count Percentages at Week 24 | Baseline, Week 24
Change from Baseline in CD4+ Cell Count Percentages at Week 48 | Baseline, Week 48
PK Parameter: Tmax of Bictegravir | Week 2 or Week 4 for Cohorts 1 & 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, & 24 hours postdose; Week 2 for Cohort 3: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, & 24 hours post-dose; Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  Tmax is defined as the time (observed time point) of Cmax. Cohorts 1 & 2 Part A will participate in an Intensive PK Evaluation at Week 2 or Week 4. Samples will be collected at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post-dose.
  Cohort 3 Part A will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose.
  Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
PK Parameter: Cmax of Bictegravir | Week 2 or Week 4 for Cohorts 1 & 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, & 24 hours postdose; Week 2 for Cohort 3: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, & 24 hours post-dose; Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  Cmax is defined as the maximum observed concentration of drug. Cohorts 1 & 2 Part A will participate in an Intensive PK Evaluation at Week 2 or Week 4. Samples will be collected at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post-dose.
  Cohort 3 Part A will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose.
  Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
PK Parameter: AUClast of Bictegravir | Week 2 or Week 4 for Cohorts 1 & 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, & 24 hours postdose; Week 2 for Cohort 3: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, & 24 hours post-dose; Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  AUClast is defined as the area under the concentration of drug from time zero to the last observable concentration. Cohorts 1 & 2 Part A will participate in an Intensive PK Evaluation at Week 2 or Week 4. Samples will be collected at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post-dose.
  Cohort 3 Part A will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose.
  Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
PK Parameter: T1/2 of Bictegravir | Week 2 or Week 4 for Cohorts 1 & 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, & 24 hours postdose; Week 2 for Cohort 3: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, & 24 hours post-dose; Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  T1/2 is defined as the estimate of the terminal elimination half-life of the drug. Cohorts 1 & 2 Part A will participate in an Intensive PK Evaluation at Week 2 or Week 4. Samples will be collected at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post-dose.
  Cohort 3 Part A will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose.
  Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
PK Parameter: Apparent Clearance (CL) of Bictegravir | Week 2 or Week 4 for Cohorts 1 & 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, & 24 hours postdose; Week 2 for Cohort 3: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, & 24 hours post-dose; Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  CL is defined as the systemic clearance of the drug following study drug administration. Cohorts 1 & 2 Part A will participate in an Intensive PK Evaluation at Week 2 or Week 4. Samples will be collected at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post-dose.
  Cohort 3 Part A will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose.
  Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
PK Parameter: Apparent Vz of Bictegravir | Week 2 or Week 4 for Cohorts 1 & 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, & 24 hours postdose; Week 2 for Cohort 3: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, & 24 hours post-dose; Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  Vz is defined as the volume of distribution of the drug after study drug administration. Cohorts 1 & 2 Part A will participate in an Intensive PK Evaluation at Week 2 or Week 4. Samples will be collected at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post-dose.
  Cohort 3 Part A will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose.
  Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
PK Parameter: AUCtau of TAF and FTC | Week 2 or Week 4 for Cohorts 1 & 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, & 24 hours postdose; Week 2 for Cohort 3: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, & 24 hours post-dose; Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval). Cohorts 1 & 2 Part A will participate in an Intensive PK Evaluation at Week 2 or Week 4. Samples will be collected at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post-dose.
  Cohort 3 Part A will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose.
  Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
PK Parameter: AUClast of TAF and FTC (Cohorts 1, 2, and 3) | Week 2 or Week 4 for Cohorts 1 & 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, & 24 hours postdose; Week 2 for Cohort 3: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, & 24 hours post-dose
  AUClast is defined as the area under the concentration of drug from time zero to the last observable concentration. Cohorts 1 & 2 Part A will participate in an Intensive PK Evaluation at Week 2 or Week 4. Samples will be collected at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post-dose.
  Cohort 3 Part A will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose.
PK Parameter: AUClast of FTC (Cohorts 4) | Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  AUClast is defined as area under the concentration versus time curve from time zero to the last quantifiable concentration.
  Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
PK Parameter: Cmax of TAF and FTC (Cohorts 1, 2, and 3) | Week 2 or Week 4 for Cohorts 1 & 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, & 24 hours postdose; Week 2 for Cohort 3: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, & 24 hours post-dose
  Cmax is defined as the maximum observed concentration of drug. Cohorts 1 & 2 Part A will participate in an Intensive PK Evaluation at Week 2 or Week 4. Samples will be collected at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post-dose.
  Cohort 3 Part A will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose.
PK Parameter: Cmax of FTC (Cohorts 4) | Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  Cmax is defined as maximum observed concentration of drug. Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
PK Parameter: Ctau of TAF and FTC | Week 2 or Week 4 for Cohorts 1 & 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, & 24 hours postdose; Week 2 for Cohort 3: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, & 24 hours post-dose; Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  Ctau is defined as the observed drug concentration at the end of the dosing interval. Cohorts 1 & 2 Part A will participate in an Intensive PK Evaluation at Week 2 or Week 4. Samples will be collected at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post-dose.
  Cohort 3 Part A will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose.
  Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
PK Parameter: Tmax of TAF and FTC | Week 2 or Week 4 for Cohorts 1 & 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, & 24 hours postdose; Week 2 for Cohort 3: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, & 24 hours post-dose; Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  Tmax is defined as the time (observed time point) of Cmax. Cohorts 1 & 2 Part A will participate in an Intensive PK Evaluation at Week 2 or Week 4. Samples will be collected at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post-dose.
  Cohort 3 Part A will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose.
  Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
PK Parameter: T1/2 of TAF and FTC | Week 2 or Week 4 for Cohorts 1 & 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, & 24 hours postdose; Week 2 for Cohort 3: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, & 24 hours post-dose; Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  T1/2 is defined as the estimate of the terminal elimination half-life of the drug. Cohorts 1 & 2 Part A will participate in an Intensive PK Evaluation at Week 2 or Week 4. Samples will be collected at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post-dose.
  Cohort 3 Part A will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose.
  Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
PK Parameter: Apparent CL of TAF and FTC | Week 2 or Week 4 for Cohorts 1 & 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, & 24 hours postdose; Week 2 for Cohort 3: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, & 24 hours post-dose; Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  CL is defined as the systemic clearance of the drug following study drug administration. Cohorts 1 & 2 Part A will participate in an Intensive PK Evaluation at Week 2 or Week 4. Samples will be collected at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post-dose.
  Cohort 3 Part A will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose.
  Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
PK Parameter: Apparent Vz of TAF and FTC | Week 2 or Week 4 for Cohorts 1 & 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, & 24 hours postdose; Week 2 for Cohort 3: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, & 24 hours post-dose; Week 2 for Cohort 4: 0 (predose) 0.5, 1, 2, 4, & 8 hours postdose
  Vz is defined as the volume of distribution of the drug after study drug administration. Cohorts 1 & 2 Part A will participate in an Intensive PK Evaluation at Week 2 or Week 4. Samples will be collected at 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post-dose.
  Cohort 3 Part A will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, and 24 hours post-dose.
  Cohort 4 Groups 2, 3, and 4 participants will participate in an Intensive PK evaluation at Week 2. Samples will be collected at 0 (pre-dose) 0.5, 1, 2, 4, and 8 hours post-dose.
Percentage of Participants Experiencing Treatment-Emergent Adverse Events Through Week 48 | Up to 48 weeks
Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities Through Week 48 | Up to 48 weeks
Acceptability of B/F/TAF Formulation at Day 1 (All Cohorts) | Day 1
  Participants or legal guardian will be asked:
  * if study drug shape and size were acceptable (for Cohort 1 and Cohort 2)
  * about ease of swallowability and the shape and size of study drug when swallowed (for Cohort 3)
  * about their understanding of instructions, preparation of the study drug formulation and study drug administration and taste (for Cohort 4)
Palatability of B/F/TAF Formulation at Day 1 (All Cohorts) | Day 1
  Participants or legal guardian will be asked about the study drug taste (All Cohorts)
Acceptability of B/F/TAF Formulation at Week 4 (All Cohorts) | Week 4
  Participants or legal guardian will be asked:
  * if study drug shape and size were acceptable (for Cohort 1 and Cohort 2)
  * about ease of swallowability and the shape and size of study drug when swallowed (for Cohort 3).
  * about their understanding of instructions, preparation of the study drug formulation and study drug administration and taste (for Cohort 4)
Palatability of B/F/TAF Formulation at Week 4 (All Cohorts) | Week 4
  Participants or legal guardian will be asked about the study drug taste (All Cohorts)
Acceptability of B/F/TAF Formulation at Week 24 (Cohort 3 and Cohort 4) | Week 24
  Participants or legal guardian will be asked:
  * about ease of swallowability and the shape and size of study drug when swallowed (for Cohort 3).
  * about their understanding of instructions, preparation of the study drug formulation and study drug administration and taste (for Cohort 4)
Palatability of B/F/TAF Formulation at Week 24 (Cohort 3 and Cohort 4) | Week 24
  Participants or legal guardian will be asked about the study drug taste
Acceptability of B/F/TAF Formulation at Week 48 (Cohort 3 and Cohort 4) | Week 48
  Participants or legal guardian will be asked:
  * about ease of swallowability and the shape and size of study drug when swallowed (for Cohort 3).
  * about their understanding of instructions, preparation of the study drug formulation and study drug administration and taste (for Cohort 4)
Palatability of B/F/TAF Formulation at Week 48 (Cohort 3 and Cohort 4) | Week 48
  Participants or legal guardian will be asked about the study drug taste
Acceptability of B/F/TAF Formulation at Week 1 (Cohort 4) | Week 1
  Participants or legal guardian will be asked about their understanding of instructions, preparation of the study drug formulation and study drug administration and taste
Palatability of B/F/TAF Formulation at Week 1 (Cohort 4) | Week 1
  Participants or legal guardian will be asked about the study drug taste
Acceptability of B/F/TAF Formulation at Week 2 (Cohort 4) | Week 2
  Participants or legal guardian will be asked about their understanding of instructions, preparation of the study drug formulation and study drug administration and taste
Palatability of B/F/TAF Formulation at Week 2 (Cohort 4) | Week 2
  Participants or legal guardian will be asked about the study drug taste

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (25):
- United States (10):
  - Children's National Health System, Washington D.C., District of Columbia
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - University of Florida Health, Gainesville, Florida
  - USF Clinic at Children's Medical Services (study visits and drug storage), Tampa, Florida
  - Grady Health System Ponce Center Family and Youth Clinic, Atlanta, Georgia
  - Wayne Pediatric Clinic, Detroit, Michigan
  - Bellevue Hospital, New York, New York
  - Duke Children's Health Center, Pediatric Infectious Diseases, Durham, North Carolina
  - St. Christopher's Hospital for Children/Section of Immunology, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- South Africa (9):
  - Department of Paediatrics and Child Health, Bloemfontein
  - Be Part Ypluntu Centre, Cape Town
  - FAMCRU, Ward J8, CapeTown
  - Dr. J Fourie Medical Centre, Dundee
  - Enhancing Care Foundation, Durban International Clinical Research Site, Durban
  - Wits RHI Shandukani Research Centre, Wits Reproductive Health & HIV Institute, Johannesburg
  - Empilweni Service and Research Unit (ESRU), Johannesburg
  - VX Pharma(Pty) Ltd, Pretoria
  - Perinatal HIV Research Unit, Soweto
- Thailand (3):
  - The HIV Netherlands Australia Thailand Research Collaboration, Bangkok
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok
  - Faculty of Medicine, Khon Kaen University, Khon Kaen
- Uganda (3):
  - Makerere University, Johns Hopkins (MU-JHU) Research Collaboration, Kampala
  - Joint Clinical Research Centre, Kampala
  - Baylor College of Medicine Children's Foundation - Uganda, Kampala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez CA, Natukunda E, Strehlau R, Venter EL, Rungmaitree S, Cunningham CK, Lalloo U, Kosalaraksa P, HellstrOm E, Liberty A, McGrath EJ, Kaur M, Leisegang R, Hindman JT, Vieira VA, Kersey K, Cotton MF, Rakhmanina N, Gaur AH. Pharmacokinetics and safety of coformulated bictegravir, emtricitabine, and tenofovir alafenamide in children aged 2 years and older with virologically suppressed HIV: a phase 2/3, open-label, single-arm study. Lancet HIV. 2024 May;11(5):e300-e308. doi: 10.1016/S2352-3018(23)00327-2. Epub 2024 Apr 12. PMID 38621393
- [Derived] Gaur AH, Cotton MF, Rodriguez CA, McGrath EJ, Helstrom E, Liberty A, Natukunda E, Kosalaraksa P, Chokephaibulkit K, Maxwell H, Wong P, Porter D, Majeed S, Yue MS, Graham H, Martin H, Brainard DM, Pikora C. Fixed-dose combination bictegravir, emtricitabine, and tenofovir alafenamide in adolescents and children with HIV: week 48 results of a single-arm, open-label, multicentre, phase 2/3 trial. Lancet Child Adolesc Health. 2021 Sep;5(9):642-651. doi: 10.1016/S2352-4642(21)00165-6. Epub 2021 Jul 22. PMID 34302760